CLINICAL TRIAL: NCT02286687
Title: Phase II Study of the PARP Inhibitor Talazoparib in Advanced Cancer Patients With Somatic Alterations in BRCA1/2, Mutations/Deletions in Other BRCA Pathway Genes and Germline Mutation in BRCA1/2 (Not Breast or Ovarian Cancer)
Brief Title: Talazoparib in Treating Patients With Recurrent, Refractory, Advanced, or Metastatic Cancers and Alterations in the BRCA Genes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2013-0961; NCI-2014-02494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0961 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-10-30; First posted 2014-11-10 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Neoplasm; ATM Gene Mutation; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Metastatic Malignant Neoplasm; PALB2 Gene Mutation; Recurrent Malignant Neoplasm; Refractory Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talazoparib) (Experimental): Patients receive talazoparib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Talazoparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase II trial studies how well talazoparib works in treating patients with cancers that have returned after a period of improvement, do not respond to treatment, or have spread to other parts of the body, and have alterations in the breast cancer, early onset (BRCA) genes. Talazoparib may cause tumor cells to die by blocking an enzyme that protects the tumor cells from damage.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the PARP inhibitor talazoparib achieves clinical benefit (complete response [CR], partial response [PR] or stable disease [SD] > 24 weeks) in metastatic or inoperable locally advanced or locally recurrent cancer patients who have somatic mutations or deletions of BRCA1 or BRCA2, mutations or homozygous deletions in other BRCA pathway genes, and germline mutations in BRCA1 or BRCA 2 with cancers other than breast or ovarian cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of talazoparib in this patient population. (Across-indication) II. To determine baseline molecular markers (deoxyribonucleic acid [DNA], ribonucleic acid [RNA] and protein) or scores (e.g., microsatellite instability positives, and somatic mutation burden) that may predict clinical benefit. (Within-indication) III. To determine pharmacodynamic (PD) markers in tumor, blood and plasma that may predict outcome. (Within-indication) IV. To determine concordance of BRCA1/2 alterations in archival tissue and pre-treatment biopsies. (Within-indication) V. To determine concordance of genomic alterations in tumor and circulating free DNA. (Within-indication) VI. To evaluate the progression free survival (PFS) in patients. (Within-indication) VII. To evaluate the duration of response (DOR) in patients. (Within-indication) VIII. To evaluate the overall survival (OR) in patients. (Within-indication)

OUTLINE:

Patients receive talazoparib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancer that is refractory to standard therapy or has relapsed after standard therapy
* Patients must have one of the following: somatic mutations or deletions in BRCA1 or BRCA2; genomic alterations in other BRCA pathway genes (subcohorts: a. ATM, b. PALB2, c. other genes, e.g. Fanconi Anemia genes, ARID1A, MER11, RAD50, NBS1, ATR; amplification of EMSY); or germline mutation in BRCA1 or BRCA 2 (not breast or ovarian cancer)
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Absolute neutrophil count >= 1500/mL
* Platelets >= 100,000/mL
* Hemoglobin >= 9 g/dL (or >= 5.6 mmol/L)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) (or glomerular filtration rate [GFR] >= 60 ml/min for patients with creatinine > 1.5 x ULN)
* Serum total bilirubin =< 1.5 x ULN (direct bilirubin =< ULN if total bilirubin [bili] > 1.5 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (or =< 5 x ULN if liver metastases [mets])
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants; activated PTT (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Patients must be >= 4 weeks beyond treatment with any chemotherapy or other investigational therapy to include hormonal, biological, or targeted agents; or at least 5 half-lives from hormonal, biological, or targeted agents, whichever is shorter at the time of treatment initiation
* Women of child-bearing potential MUST have a negative serum or urine human chorionic gonadotropin (HCG) test unless prior tubal ligation (>= 1 year before screening), total hysterectomy or menopause (defined as 12 consecutive months of amenorrhea); patients should not become pregnant or breastfeed while on this study; sexually active patients must agree to use dual contraception for the duration of study participation and for 120 days after the last dose of talazoparib
* Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures
* Patients need to have biopsiable disease to enroll on cohort 1-2; patients eligible for cohort 3 with a germline BRCA alteration can be enrolled even if they do not have biopsiable disease

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Prior treatment with a PARP inhibitor
* Known hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Inability or unwillingness to swallow pills
* Active infection requiring intravenous (IV) antibiotics or other uncontrolled intercurrent illness requiring hospitalization
* Any medical condition or diagnosis that would likely impair absorption of an orally administered drug (e.g. gastrectomy, ileal bypass, chronic diarrhea, gastroparesis)
* Inability to comply with the study and follow-up procedures
* History of cerebrovascular accident (CVA), myocardial infarction or unstable angina within the previous 6 months before starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless or clinical stability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-12-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit by Response Evaluation Criteria in Solid Tumors 1.1 | Up to 1 year
  Evaluated separately in each cohort. Calculated using posterior probabilities along with corresponding credible intervals.

SECONDARY OUTCOMES:
Progression free survival | Up to 1 year
  Calculated using the Kaplan-Meier method.
Overall survival | Up to 1 year
  Calculated using the Kaplan-Meier method.
Duration of response | Up to 1 year
  Calculated using the Kaplan-Meier method.

OTHER OUTCOMES:
Molecular markers that may predict clinical benefit | Baseline
  Marker values will be compared between patients with and without clinical benefit using chi-squared or Fisher exact tests for categorically-scaled markers and Wilcoxon rank sum tests for interval- and ordinal-scaled markers. Only those significant on univariate analysis will be combined into a single logistic regression model to assess their independent effects on clinical benefit. Analyses will be performed both within and across the five cohorts.
Pharmacodynamic markers in blood and plasma that may predict outcome | Up to week 4
  Regulation of poly-adenosine triphosphate ribose activity in peripheral blood mononuclear cells will be correlated with response. Effect of treatment on proteomic profile and cell-free deoxyribonucleic acid will be assessed as exploratory endpoints.
BRCA1/2 alterations in archival tissue | Baseline
  Concordance between archival tissue and pre-treatment biopsies will be assessed using kappa statistics.
BRCA1/2 alterations in pretreatment biopsies | Baseline
  Concordance between archival tissue and pre-treatment biopsies will be assessed using kappa statistics.
Genomic alterations in tumor deoxyribonucleic acid | Baseline
  Concordance between tumor and circulating free deoxyribonucleic acid will be assessed using kappa statistics.
Genomic alterations in circulating free deoxyribonucleic acid | Up to week 4
  Concordance between tumor and circulating free deoxyribonucleic acid will be assessed using kappa statistics.
Change in marker levels | Baseline to 2 weeks
  The markers described yield interval-scaled values that may not be normally distributed, so differences between baseline and 2-week values will be assessed using the Wilcoxon signed-rank test.
Baseline proteomic signature and pharmacodynamic response by reverse phase protein array | Baseline
  Pharmacodynamic effect of talazoparib on proteomic signature will be assessed by reverse phase protein array and correlated with response, clinical benefit, as well as best response as percentage tumor change.
Archival immunohistochemistry staining | Baseline
  Immunohistochemistry staining will be assessed via the H-score which can be treated as an interval-scaled variable. The concordance correlation coefficient as well as the Altman-Bland approach will be used to assess the concordance between archival immunohistochemistry staining and baseline biopsy immunohistochemistry staining. In addition, PTEN will be assessed (PTEN loss, no loss). Concordance between archival tissue and pre-treatment biopsies will be assessed using kappa statistics.
Baseline biopsy immunohistochemistry staining | Baseline
  Immunohistochemistry staining will be assessed via the H-score which can be treated as an interval-scaled variable. The concordance correlation coefficient as well as the Altman-Bland approach will be used to assess the concordance between archival immunohistochemistry staining and baseline biopsy immunohistochemistry staining. In addition, PTEN will be assessed (PTEN loss, no loss). Concordance between archival tissue and pre-treatment biopsies will be assessed using kappa statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A Piha-Paul, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org